CLINICAL TRIAL: NCT01497483
Title: The Pharmacokinetic Interaction Between Pravastatin and Cyclosporine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study With Pravastatin and Cyclosporine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 11-06315; U01GM061390 (NIH)
Record Dates: First submitted 2011-12-07; First posted 2011-12-22 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — Pravastatin; Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pravastatin alone (Active Comparator): Subjects will be dosed with Pravastatin alone (40 mg)
  Interventions: Drug: Pravastatin alone
- Pravastatin and Cyclosporine (Experimental): Subjects will be dosed with pravastatin and cyclosporine.
  Interventions: Drug: Pravastatin and Cyclosporine

INTERVENTIONS:
Drug: Pravastatin alone — Pravastatin 40 mg with placebo.
  Arms: Pravastatin alone
Drug: Pravastatin and Cyclosporine — Pravastatin 40 mg co-administered with 200 mg of cyclosporine.
  Arms: Pravastatin and Cyclosporine

SUMMARY:
This study will address the following question: Does cyclosporine affect the pharmacokinetics of pravastatin in healthy volunteers? Studies have shown that cyclosporine inhibits the organic anion transporter required for pravastatin transport into the liver, thus increasing pravastatin levels in the blood. The investigators hypothesize that this inhibition will vary among people based on genetic differences. This knowledge is important to help develop safer and more effective drug therapy with reduced side effects.

DETAILED DESCRIPTION:
Screening Procedures:

Prior to enrollment, subjects will be asked to come to the Clinical and Translational Science (CTSI) Clinical Research Center (CRC) at San Francisco General Hospital (SFGH). The study protocol and procedures will be explained in detail, all questions will be answered, and subjects will be provided with a consent form to sign. The screening visit will be conducted within 14 days of the first inpatient visit (i.e. first pravastatin with placebo or pravastatin with cyclosporine dosing day)

Only after subjects have consented to participate in the study will the screening procedures commence. During the screening visit, vital signs as well as blood sample (10 mL) will be taken by venipuncture to measure a complete blood count (CBC), electrolytes, blood urea nitrogen (BUN), creatinine, and liver function tests (LFTs) to screen for anemia and renal or hepatic insufficiency (see Inclusion/Exclusion Criteria)

Procedures During Main Study:

An equal number of subjects will be randomized, by a computer program, into one of the two study arms described below. On the first day of the study, subjects will be dosed with either 100 mg cyclosporine or placebo at 8PM, followed by an overnight fast. On the morning of Day 2, subjects will be asked to take a second dose of 100 mg cyclosporine or placebo at 8AM. At 9AM of Day 2, subjects will be asked to take 40 mg pravastatin. Plasma samples (5 ml) will be collected at baseline (prior to pravastatin administration), then at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12 hours post-dose. Whole blood will also be collected 12 hours post-dose to measure the cyclosporine level.

The procedures during the second visit of the study will be identical to the first, but with dosing of 100 mg cyclosporine or placebo, opposite of what was dosed at the first study visit.

Clinical and Laboratory Determinations:

Analytical Methods:

Measurement of pravastatin in plasma will be performed by High Performance Liquid Chromatography (HPLC) with tandem mass spectrometry (MS/MS), using assays previously described and validated.

ELIGIBILITY:
Inclusion Criteria:

* Carrier of one of the three SLCO1B1 polymorphisms that we are studying (SLCO1B1 521TT, 521TC, 521CC)
* Men or women (women must have negative pregnancy test)
* ages 18 to 45 years
* Caucasian
* Healthy, including no renal or hepatic disease, as determined from plasma creatinine and liver enzyme levels
* No medications currently, except for vitamins and oral contraceptive pills
* Willingness to spend two nights at the San Francisco General Hospital
* Sign informed consent

Exclusion Criteria:

* Under 18 years old
* Unable to confirm Caucasian ancestry
* Pregnant or lactating women (female subjects will have a urine pregnancy test at the screening visit)
* Prior history of allergic reaction to pravastatin or cyclosporine
* Has a risk of congestive heart failure requiring pharmacologic treatment (medical history)
* Has prior renal or hepatic dysfunction
* Risk of urinary or gastric retention or narrow-angle glaucoma (by medical history examination)
* Impaired renal function (e.g. as suggested by abnormal creatinine clearance, eGFR < 60 or serum creatinine > 1.4 mg/dl in females and > 1.5 mg/dl in males) which may also result from conditions such as cardiovascular collapse (shock), acute myocardial infarction (heart attack), and septicemia, abnormal heart rhythms (tachyarrhythmias; heart beat > 100 beats per minute)
* Impaired hepatic function (> 1.5 times the upper limit of normal)
* Evidence of anemia (hemoglobin <10g)
* Taking medications other than vitamins that could confound study results
* They do not provide informed consent to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics of co-administration of pravastatin & cyclosporine in healthy volunteers | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Kroetz, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hosptail, San Francisco, California, United States